CLINICAL TRIAL: NCT00255112
Title: Psychological Treatment of Separation Anxiety Disorder
Brief Title: TAFF-Psychological Treatment of Separation Anxiety Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Swiss National Science Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PP001--68701; Trennungsangstprojekt NZX 1303
Record Dates: First submitted 2005-11-16; First posted 2005-11-17 (Estimated); Last update posted 2015-06-11 (Estimated); Status verified 2015-06

CONDITIONS: Separation Anxiety Disorder
Keywords: SAD; treatment; cognitive behavior therapy; family; children; anxiety
MeSH Terms: conditions — Anxiety, Separation; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (No Intervention): The present study evaluates the efficacy of a family-based CBT treatment specifically tailored to children with SAD, developed at the University of Basel. The study consists of 40 participants (5-7 years old) with SAD and their families. Participants were randomly assigned to 12 weeks of SAD-specific family-based CBT treatment or to waitlist condition.
- 2 (Active Comparator): The present study evaluates the efficacy of a family-based CBT treatment specifically tailored to children with SAD, developed at the University of Basel in comparison to a global CBT treatment. The study consists of 60 participants (between 8 and 13 years old), randomly assigned to one of the two treatments.
  Interventions: Behavioral: family based cognitive behavior therapy

INTERVENTIONS:
Behavioral: family based cognitive behavior therapy — newly developed family based cognitive behavior therapy for children with separation anxiety disorder over 5 years old
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether a specific family based cognitive behavioral treatment program is effective in the treatment of children with separation anxiety disorder.

DETAILED DESCRIPTION:
Anxiety disorders are the most common mental disorders both in adulthood and childhood. Recent research indicates that anxiety disorders in childhood and in particular Separation Anxiety Disorder (SAD) increase the risk of mental disorders in adulthood. Despite these results research on SAD is still limited compared to the vast research activity on adult anxiety disorders. The proposed research program will close a gap of current international research: It will test the efficacy of a family based cognitive behavioral treatment program specific for SAD.

The research program consists of two parts. One study is aimed at children with SAD aged 5 to 7. 40 children are randomly allocated immediately to SAD-specific family-based treatment or to a wait list. For the second study 60 children with SAD (8 to 13 years old) are randomly allocated to either SAD-specific family-based treatment ("SAD-CBT") or a well established global CBT program for childhood anxiety disorders ("global CBT").

In both studies treatment success is tested at the end of treatment as well as 4 weeks and 1, 2 and 3 years after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of SAD
* Age 5 to 13 years
* Knowledge of German language
* Consent to randomization and psychological testing

Exclusion Criteria:

* Comorbid Pervasive Developmental Disorders
* Active psychotropic drugs

Ages: 5 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2004-06; Primary Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
DSM-IV criteria for Separation Anxiety Disorder | December 2009
Global Success Rating (GSR) | December 2009
Separation Anxiety Inventory for Children (SAI) | December 2009

SECONDARY OUTCOMES:
Revised Children's Manifest Anxiety Scale (RCMAS) | December 2009
Sheehan Disability Scale (SDS) | December 2009
Inventory for the Assessment of Quality of Life in Children and Adolescents (IQL) | December 2009

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Schneider, Prof. Dr., Study Chair — Ruhr-Universität, Bochum, Germany
Locations (1):
- Institute of Psychology, Basel, Canton of Basel-City, Switzerland

REFERENCES:
- [Derived] Schneider S, Blatter-Meunier J, Herren C, Adornetto C, In-Albon T, Lavallee K. Disorder-specific cognitive-behavioral therapy for separation anxiety disorder in young children: a randomized waiting-list-controlled trial. Psychother Psychosom. 2011;80(4):206-15. doi: 10.1159/000323444. Epub 2011 Apr 14. PMID 21494062
- See also: Related Info — http://www.taff.unibas.ch